CLINICAL TRIAL: NCT02733731
Title: The Treatment Effect of Chinese Herbal Compound Ointment on Atrophic Vaginitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhou Xin, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Zxin
Record Dates: First submitted 2016-03-20; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Estriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Chinese Herbal Compound Ointment (Experimental): This kind of CHCO composed of several chinese herbs,dong quai,angelica,resina draconis and lithospermum.The dosage of medicine for single treatment once a day in two group is 0.5g,The total time for therapy is 3 weeks.
  Interventions: Drug: Chinese Herbal Compound Ointment
- Estriol (Active Comparator): The dosage of medicine for single treatment once a day in two group is 0.5g,The total time for therapy is 3 weeks in two groups.
  Interventions: Drug: Estriol

INTERVENTIONS:
Drug: Chinese Herbal Compound Ointment
  Arms: Chinese Herbal Compound Ointment
Drug: Estriol
  Arms: Estriol

SUMMARY:
Objective：To evaluate the effect and safety of the traditional chinese medicine oil agent on senile atrophic compared as compared to estriol cream in aged woman.

Design: A randomized double-blind controlled trial.

Setting: The hospital ward.

Participants: 200 postmenopausal woman with senile vaginitis (mean age 56).

Intervention: The traditional chinese medicine oil and estriol cream were separately intravaginal administrated in treatment group and control group for 3 weeks，follow-up 1 month.

Measurement: symptom improving(pain and itch) and onset time, edema-size of vaginal wall, vaginal discharge, and PH changes.

DETAILED DESCRIPTION:
80 postmenopausal women living in the communities near the hospital with AV (atrophic vaginitis) symptoms were recruited for this clinical trial. Patients with AV receiving external treatment and requiring hospitalization were randomized in a double-blind, single-centre trial. Subjects received CHCO (Chinese Herbal Compound Ointment) topical vaginal application in experimental group, while estriol in control group. The dosage of medicine for single treatment once a day in two group is 0.5g.The total time for therapy is 3 weeks in two groups. Assessment indicators：vagine PH, sIgA and IL-1βchanges, the degree of symptoms improving, onset time, edema-size of vaginal wall, vaginal discharge, and relapses and retreatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* With typical clinical manifestations: virginal genital itching or burning sense, Increased vaginal secretions, a yellow, a serious bloody pus-like leucorrhea, or sexual intercourse pain
* Gynecological examination: Vaginal epithelium atrophy，Vaginal folds flat or disappear， mucosal hyperemia， superficial ulceration
* Both ALT and AST are normal or less than 2 times, bilirubin is normal
* Serum creatinine level is within the normal range
* ECG is normal;

Exclusion Criteria:

* Gynecological and breast Oncology, endometrial hyperplasia(≥5mm)
* Estrogenic drugs or probiotics used in four week
* Participate in other clinical trials;Thrombotic diseases
* Abnormal vaginal bleeding without clear diagnose
* Estriol allergy
* Severe pneumonia, tuberculosis, lung abscess, myocarditis
* heart,liver or kidney failure(NYHA class III-IV,ALT to AST ratio twice more than upper limit of normal
* sexually transmitted diseases;mental disorders

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
symptom questionnaire scores | 77days
sign questionnaire scores | 77days

SECONDARY OUTCOMES:
recurrence rate retreatment effect | Within 28days after treatment
retreatment effective rate | Within 56days after treatment
PH value of vaginae secretion | 49days
sIgA value of vaginae secretion | 49days
IL-1βvalue of vaginae secretion | 49days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun-yat Sen University, Guangzhou, Guangdong, China